CLINICAL TRIAL: NCT05054647
Title: Mental Stress Symptoms in Family Caregivers of Palliative Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 33-332; 33-332 (Other: Ethikkommission Medizinische Universität Graz)
Record Dates: First submitted 2021-06-30; First posted 2021-09-23 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Family Caregivers; Palliative Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- family caregivers of palliative patients: psychometric questionnaires
  Interventions: Other: psychometric questionnaires

INTERVENTIONS:
Other: psychometric questionnaires — Perceived Stress Scale (PSS-10); Trier-Inventory on Chronic Stress; State/Trait Anxiety Inventory (STAI); AVEM-Work-related behaviour and experience pattern; Maslach Burn-out Inventory - Human Services Survey (MBI - HSS) health-related anxiety: Whiteley Index (WI)

SUMMARY:
Receiving a life-limiting diagnosis is often a shock for those affected as well as for their relatives, which changes the entire life situation of the family. New perspectives often arise, as well as feelings of worry, sadness and powerlessness. Caregiving is often an extreme physical challenge, but above all a psychological one.

Aims of the study

1. To investigate whether family caregivers of palliative patients with severe trait anxiety in the care situation also suffer from severe state anxiety.
2. To investigate whether family caregivers of palliative patients with increased stress levels and burnout-promoting work-related behaviour suffer more from burnout symptoms, health-related anxiety and psychosomatic complaints.
3. To investigate the impact of nursing support by a mobile palliative team on family caregivers of palliative patients.

ELIGIBILITY:
Inclusion criteria:

* Women and men between 18 and 90 years of age
* Current palliative care situation of a relative with a life-limiting diagnosis.

Exclusion criteria:

* Persons incapable of giving consent (e.g. dementia, delirium, etc.)
* Failure to meet the inclusion criteria

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Family caregivers of palliative patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
burn-out syndrome, Outcome is the difference between measurement 1 (Baseline) and measurement 2 (Follow-up) | 2 months
  Maslach Burn-out Inventory (MBI), The MBI does not provide a single score but a profile.

SECONDARY OUTCOMES:
health-related anxiety, Outcome is the difference between measurement 1 (Baseline) and measurement 2 (Follow-up) | 2 months
  Whiteley Index/Illness Attitude Scale (WI-IAS). Whitely-Index: The Whitely-Index is formed by the sum of the points for each answer - the higher the score, the more likely one is to be hypochondriacal.
  IAS: The total score ranges from 0 to108.
State/Trait anxiety, Outcome is the difference between measurement 1 (Baseline) and measurement 2 (Follow-up) | 2 months
  State-Trait Anxiety Inventory (STAI). Scores range from 20 to 80, with higher scores correlating with greater anxiety.
Work-related behaviour and experience pattern, Outcome is the difference between measurement 1 (Baseline) and measurement 2. | 2 months
  Work-related behaviour and experience pattern (AVEM), The AVEM questionnaire does not provide a single score but a profile.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Baranyi, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided